CLINICAL TRIAL: NCT04955340
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, Excretion of [14C]-Resminostat Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Phase 1, Open-label Study of the Absorption, Metabolism, Excretion of [14C]-Resminostat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 4SC AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4SC-201-7-2020; 2021-000555-39 (EudraCT Number); 8448213 (Other: Covance Study Number)
Record Dates: First submitted 2021-06-23; First posted 2021-07-08 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Cutaneous T Cell Lymphoma; Mycosis Fungoides; Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]-resminostat (Experimental): single dose of 400 mg [14C]-resminostat
  Interventions: Drug: [14C]-resminostat

INTERVENTIONS:
Drug: [14C]-resminostat — 1 single dose of 400 mg [14C]-resminostat

SUMMARY:
Resminostat is a potent, orally available inhibitor of Class I, IIb and IV histone deacetylases (HDACs), including a pronounced activity against HDAC6. Resminostat targets epigenetic changes observed in tumour cells and has the potential to provide significant benefit to patients with advanced malignancies by inhibiting tumour progression and metastasis or even inducing tumour regression.

This will be a Phase 1, open-label, non-randomized, single dose study of the absorption, metabolism, excretion of [14C] resminostat following a single oral dose in healthy male participants.

The purpose of this study is to determine the absorption, metabolism, and excretion (AME) of [14C] resminostat and to characterize and determine the metabolites present in plasma, urine, and, where possible, faeces in healthy male participants following a single oral administration. Knowledge of the metabolism and excretion of parent drug and its metabolites is useful for evaluating the Metabolites in Safety Testing requirements elucidated in the International Conference on Harmonisation (ICH) M3, and the likelihood of effects of renal or hepatic impairment on the disposition of resminostat, and the likelihood for drug-drug interactions with resminostat. The results from this study may guide future study designs using special populations or evaluating the potential for drug-drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 35 (inclusive) and 55 years of age (inclusive)
* Body mass index between 18.0 and 28.0 kg/m2, inclusive but at least 60 kg of body weight.
* Healthy, as determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert Meulengracht's syndrome based on total and direct bilirubin] is not acceptable) at screening and/or check-in as assessed by the investigator (or designee).
* Subjects must agree to use contraception
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions
* History of a minimum of 1 bowel movement per day.
* Subjects must agree not to donate sperm from check-in until 90 days after discharge.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* Any of the following abnormalities in laboratory test values and/or ECG at screening and/or check-in, confirmed by repeat: hemoglobin, white blood cell count, total platelets, and QTcF outside of normal range; alanine aminotransferase, aspartate aminotransferase, and creatinine values > upper limit of normal; and estimated glomerular filtration rate (calculated using Cockcroft-Gault formula) <60 mL/min.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
* Confirmed (eg, 2 consecutive measurements) systolic blood pressure >150 or <90 mmHg, diastolic blood pressure >90 or <50 mmHg, and pulse rate >90 or <40 beats per minute.
* History of alcoholism or drug/chemical abuse within 2 years prior to screening.
* Alcohol consumption of > 21 units per week. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
* Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at screening or check-in.
* Positive hepatitis panel and/or positive human immunodeficiency virus test
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days or 5 half-lives, whichever is longer prior to dosing.
* Administration of any vaccination (including vaccines currently being deployed in the UK for SARS-CoV-27) within the past 90 days prior to dosing.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, and excretion processes, including St. John's wort, within 30 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use any prescription medications/products within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use of tobacco- or nicotine-containing products within 3 months prior to check-in, or positive cotinine test at screening or check-in.
* Ingestion of poppy seed-, Seville orange-, or grapefruit-containing foods or beverages within 7 days prior to check-in.
* Receipt of blood products within 2 months prior to check-in.
* Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
* Poor peripheral venous access
* Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
* Subjects who have participated in any clinical study involving a radiolabeled investigational product within 12 months prior to check-in.
* Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
AUC0-tlast | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  AUC from time zero to the last quantifiable concentration derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
AUC0-∞ | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  AUC from time zero extrapolated to infinity derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
Cmax | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  maximum observed concentration derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
tmax | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  time to reach Cmax derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
tlag | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  time to the first quantifiable concentration in plasma derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
λz | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  terminal elimination rate constant derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
t1/2 | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  apparent terminal elimination half-life derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
CL/F | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  apparent total clearance derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
Vz/F | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  apparent volume of distribution derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
AUC0-∞ Plasma resminostat/Total Radioactivity Ratio | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  AUC0-∞ of plasma resminostat relative to AUC0-∞ of plasma total radioactivity derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
AUC0-∞ Blood/Plasma Ratio | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  AUC0-∞ of whole blood total radioactivity to AUC0-∞ of plasma total radioactivity derived from the whole blood and plasma concentration-time profiles following oral administration of [14C]-resminostat
Aeu | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  amount excreted in urine derived from urine collections at each sampling interval
cumulative Aeu | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  cumulative amount excreted in urine derived from urine collections at each sampling interval
feu | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  percentage excreted in urine derived from urine collections at each sampling interval
cumulative feu | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  cumulative percentage excreted in urine derived from urine collections at each sampling interval
Aef | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  amount excreted in feces derived from feces collections at each sampling interval
cumulative Aef | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  cumulative amount excreted in feces derived from feces collections at each sampling interval
fef | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  percentage excreted in feces derived from feces collections at each sampling interval
cumulative fef. | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  cumulative percentage excreted in feces derived from feces collections at each sampling interval

SECONDARY OUTCOMES:
Safety and Tolerability | from study drug intake until 28 days after study drug administration
  AE reporting including relatedness and severity
Heart rhythm | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  ECG analysis by 12-lead ECG
Ventricular rate | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  ECG analysis by 12-lead ECG
PR-interval (synonymous: PQ interval) | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  ECG analysis by 12-lead ECG
QRS complex | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  ECG analysis by 12-lead ECG
QT interval | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  ECG analysis by 12-lead ECG
QTcF interval | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  ECG analysis by 12-lead ECG
Vital Signs (Body Temperature) | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  Body temperature will be measured after a 5 minute rest in supine position
Vital Signs (Blood pressure) | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  Systolic and diastolic blood pressure will be measured after a 5 minute rest in supine position
Physical Examination | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  A full physical examination covering at least head, eyes, ears, nose and throat, lungs, heart, neurological status, abdomen, extremities, skin, and lymph nodes
metabolic profiles of resminostat | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  identification and quantification of metabolites in serum and urin samples by HPLC
identification and quantification of resminostat metabolites | From day -1 until maximum 15 days after single dose of [14C]-resminostat
  identification and quantification of metabolites in serum and urin samples by HPLC

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical research Unit Ltd., Leeds, United Kingdom